CLINICAL TRIAL: NCT04055272
Title: A Mobile Text Messaging Intervention for Indoor Tanning Addiction
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Georgetown University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: STUDY00000474
Record Dates: First submitted 2019-08-01; First posted 2019-08-13 (Actual); Last update posted 2022-08-04 (Actual); Status verified 2022-07

CONDITIONS: Indoor Tanning
Keywords: indoor tanning; skin cancer; mobile health; text messaging
MeSH Terms: conditions — Skin Neoplasms

STUDY DESIGN:
Intervention Model Description: This is a randomized trial with two groups: 1) Indoor tanning education only; 2) Mobile text messaging intervention
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Text messaging (Experimental): Participants in the text messaging intervention arm receive mobile text messages communicating the risks of indoor tanning and motivating cessation on their mobile phones
  Interventions: Behavioral: Mobile text messaging intervention
- Control (No Intervention): Participants in the control arm receive no intervention

INTERVENTIONS:
Behavioral: Mobile text messaging intervention — Participants in the intervention arm will receive text messages to their mobile phones designed to communicate the risks of indoor tanning and motivate cessation. The intervention exposure lasts for 4 weeks with messages sent 2 days each week. It is an interactive intervention that engages participants by asking them to respond to prompts, and sending indoor tanning message content in return on message days.
  Arms: Text messaging

SUMMARY:
The purpose of this study is to test the effects of messages communicating the risks (i.e., health harms, addictiveness) of indoor tanning delivered via mobile text messaging among young adult women ages 18 to 30 years who meet screening criteria for indoor tanning addiction.

DETAILED DESCRIPTION:
This is a two arm randomized controlled trial to test the effects of messages communicating the risks of indoor tanning delivered via mobile text messaging as a strategy for promoting cessation among young adult women who meet screening criteria for indoor tanning addiction. Eligible participants are young adult women ages 18 to 30 years who meet screening criteria for indoor tanning addiction and have access to the internet and a personal mobile phone to complete study procedures. Participants will complete baseline measures and then be randomized to the study arms. The text messaging intervention exposure in the intervention arm will last for four weeks. The control arm will be given basic indoor tanning education information and will not receive any intervention. Follow up assessments capturing study outcomes will be administered at 1 month (i.e., immediately post-intervention) and three months post-intervention.

ELIGIBILITY:
Inclusion Criteria:

* Female
* Age between 18 and 30 years
* Meet self-report criteria for tanning addiction
* Has access to the internet to complete study procedures
* Has personal mobile phone to complete study procedures

Exclusion Criteria:

* Male
* Age less than 18 or greater than 30
* Does not meet self-report criteria for tanning addiction
* Does not have access to the internet to complete study procedures
* Does not have a personal mobile phone to complete study procedures

Ages: 18 Years to 30 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 265 (Actual)
Dates: Start 2020-01-07 (Actual); Primary Completion 2022-03-31 (Actual); Study Completion 2022-03-31 (Actual)

PRIMARY OUTCOMES:
Motivation to Quit Indoor Tanning | 1 month follow up
  Motivation to quit is measured by participant report by a single question with a 1 to 7 response scale. Higher scores indicate greater motivation to quit and are considered better outcomes. This question is administered at 1 month follow up and at 3 month follow up.
Indoor Tanning Cessation | 1 month follow up
  Indoor tanning cessation is measured by participant report by a single question asking if participants have stopped indoor tanning completely. Responses indicating cessation are considered better outcomes. This item is administered at 1-month follow-up and at 3 month follow up.

SECONDARY OUTCOMES:
Attempts to Quit Indoor Tanning | 1 month follow up and 3 month follow up
  Attempts to quit indoor tanning are measured by participant report by a single question asking if participants have attempted to quit indoor tanning since the last assessment. Responses indicating any attempt(s) to quit are considered a better outcome. This item is administered at 1 month follow up and at 3 month follow up.

OTHER OUTCOMES:
Risk Appraisals | 1 month follow up and 3 month follow up
  Perceived risk of harm are measured by asking participants how likely harms are to occur (1 = no chance, 7 = certain to happen). Worry about harms are measured by asking participants how worried they are about harms of indoor tanning (1 = not at all, 7 = very much). Greater risk appraisals are considered a better outcome. The items are administered at 1 month follow up and at 3 month follow up.
Efficacy Beliefs | 1 month follow up and 3 month follow up
  Beliefs about the health benefits of quitting indoor tanning, efficacy beliefs, are measured using 6 questions asking about health benefits occurring from quitting indoor tanning (1 = No Chance, 7 = Certain to Happen). Greater efficacy beliefs are considered a better outcome. These items are administered at 1 month follow up and at 3 month follow up.

CONTACTS AND LOCATIONS:
Overall Officials: Darren Mays, PhD, MPH, Principal Investigator — Georgetown University
Locations (1):
- Georgetown University, Washington D.C., District of Columbia, United States

IPD SHARING:
Plan to Share IPD: Undecided
We will consider requests to share de-identified IPD individually and according to the investigator's study protocol and institutional data sharing policy.